CLINICAL TRIAL: NCT06118879
Title: Role of Sensory Deficits and the Effect of Sensory Stimulation on Sensorimotor Control and Neuromuscular Performance in Athletes With Chronic Ankle Instability
Brief Title: Role of Sensory Deficits on Sensorimotor Control in Athletes With Chronic Ankle Instability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NYCU112052AF
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Chronic Ankle Instability
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sensory level stimulation with exercise (Experimental)
  Interventions: Device: Transcutaneous electrical stimulation
- Sham stimulation with exercise (Sham Comparator)
  Interventions: Device: Transcutaneous electrical stimulation
- Exercsie alone (Active Comparator)
  Interventions: Device: Transcutaneous electrical stimulation

INTERVENTIONS:
Device: Transcutaneous electrical stimulation — sensory level stimulation, one-leg standing and Y-balance training
  Other Names: Neuromuscular training exercise

SUMMARY:
Purpose: Chronic ankle instability (CAI), characterized by instances of repetitive sprains and giving way, is a common chronic dysfunction among athletes. Despite well documented evidence showing impaired peripheral sensory and both central and peripheral motor control, little was known regarding how CAI affects somatosensory cortical activation. Traditionally, management of CAI mostly focused on restoration of motor deficits, with less emphasis on sensory pathway deficits. Only few sensory targeted intervention methods including joint mobilization and massage, have been described. However, methods such as joint mobilization provide not only sensory stimulation but also mechanical alignment correction. In addition, these studies showed functional improvement without exploring mechanisms. Therefore we would like to apply for a three year study grant to firstly investigate the effect of CAI on peripheral and central somatosensation and neuromuscular performance; and secondly to examine the immediate effect of sensory-level electrical stimulation on neurophysiological variables and neuromuscular performance; and lastly to determine the short-term effect of intervention (sensory stimulation with exercise, sham stimulation with exercise, and exercise alone) in athletes with CAI.

Research design and methods: This is a cross-sectional exploratory and randomized controlled study. For the first year, we plan to recruit 45 young athletes (20-40 years old) with CAI and 15 matched controls to compare the somatosensory evoked potentials (SEPs), corticomuscular coherence (CMC), α- band event-related desynchronization (ERD), proprioception, two point discrimination threshold of the plantar surfaces, muscle activation and reaching distances of the Y balance test. Activity in the sensorimotor cortex will be recorded using a 64-chanel EEG (SAGA 32/64+ for EEG). Muscle activation is measured using an 8-channel electromyography (EMG) system (Noraxon myo METRICS Portable Lab, Noraxon U.S.A.). For the second year, the 45 young adults with CAI will be randomized into the sensory stimulation (TENS) group, the sham stimulation group, or the control group. The TENS group will receive 40 minutes of sensory electrical stimulation, and the sham group will receive 30 seconds of sensory stimulation at the beginning and end of the treatment. The control group will rest for 40 minutes. The assessment items are identical to those in the first year, and will be carried out before and immediately after the intervention. For the third year, the 45 young adults with CAI will be randomized into the exercise with sensory stimulation (EX-TENS) group, exercise with sham stimulation (EX-ss) group, or exercise alone (EX) group. Participants will receive five sessions of intervention (30 minutes neuromuscular training with or without 40 min stimulation) within two weeks and the assessment will be carried out before and after the intervention.

Data analysis: Comparisons of all continuous variables are performed using oneway analysis of variance (ANOVA), and repeated measures ANOVA. The significance level is set at 0.05. Significance.

Results of this study provide a better understanding for central somatosensory control mechanisms for chronic ankle instability, and help clinicians and trainers to choose the most appropriate training strategy for people with unstable ankles. We plan to present our work in 3-4 international conferences, and publish 2-3 papers in SCI journals in 5 years.

DETAILED DESCRIPTION:
Characteristics of the chronic ankle instability (CAI): Lateral ankle sprain is one of the most common musculoskeletal injuries in the sports clinics. The high prevalence of lateral ankle sprains, combined with a high recurrence rate and persistent post sprain symptoms make lateral ankle sprains and their sequelae a significant health impact and healthcare burden. Although lateral ankle sprains are generally considered benign injuries, it is estimated that 40% of individuals with lateral ankle sprains will subsequently develop chronic ankle instability within the first year after a lateral ankle sprain.

Chronic ankle instability is characterized by repetitive sprains, perceived instability, and giving way, which can be classified into two categories: mechanical and functional ankle instability. Mechanical instability of the ankle is a result of loss of mechanical structural constraints (i.e., ligaments); whereas functional instability refers to instability related to altered postural control and reduced functional capacity due to impaired sensorimotor control including altered muscle recruitment around the ankle and impairment of the proprioceptive system etc.. In addition to interfering with sporting performance, and CAI has been found to be associated with lower quality of life and increased likelihood (68%-75%) of developing ankle arthritis. Hertel reported that individuals with ankle instability had higher risk of recurrent ankle sprains, and the treatment for symptoms of CAI could be time-consuming and costly. Numerous impairments have been reported associated with CAI, ranging from loss of joint mobility and muscle strength, compromised proprioception and sensation, poor postural control and neuromuscular performance, and altered movement patterns. However, the mechanisms and management strategies are still not clearly understood in many aspects. And thus, a great variety of intervention has been proposed with inconsistent results reported.

Conceptual model for the development of CAI: The theory linking poor neuromuscular control and CAI has been discussed for more than half a century. It was believed that after the ankle sprain, some of the joint receptors and peripheral nerve fibers around the ankle joint were affected, resulting in impaired reflex responses and functional stability of the ankle. More researchers later reported that CAI not only presented with sensory deficits, but also deficits in motor control, and these changes in sensorimotor system would eventually lead to loss of function. In 2019, Hertel et al. (2019) revised the current model for the development of CAI. It is proposed that the initial ankle injury would influence the neural system, disturbing the balance and stability between the sensation, perception and motor function. These disturbances would lead to self-adjustment of the sensorimotor system to attempt to adapt to the altered condition, and consequently might result in long term changes in neural network, and expose individuals to persistent symptoms of instability. This newly revised model integrates both peripheral and central sensorimotor systems to explain the development of CAI; but it clearly shows that the central sensorimotor processing in individuals with CAI is less explored, particularly for the impact of CAI on the somatosensory cortex.

Individuals with CAI have poorer neuromuscular performance: The effect of CAI on the neuromuscular control and posture stability has been extensively studied. The research topics of interest included altered reflexes and neuromuscular inhibition, muscle activation patterns (timing, recruitment order, and amplitude) and joint mechanics of the lower extremity segments during sudden inversion perturbation or jump landing, and posture control characteristics during balance testing tasks. It is generally agreed that people with CAI had lower Hmax/Mmax ratios (H reflex/M reflex ratios) of the soleus and peroneus longus muscle than those un-injured controls, indicating that neural excitability of the spinal level in those with CAI was depressed; this population also presented with altered muscle activation of the peroneus, tibialis anterior and soleus muscles, and changed balance control strategies. Recent publications of systematic review and meta-analysis by Hoch and McKeon (2014) and by Thompson et al. (2018) showed that there was a strong evidence to support dynamic balance, peroneal reaction, and eversion strength deficits contributing to CAI. Because of the strong evidence showing motor impairment in CAI, the dominant intervention strategy for this population has been motor performance driven so far.

Deficits in somatosensation in people with CAI Proprioceptive deficits in CAI have been the main focus of research for decades. Thompsons et al. (2018) indicated that there was moderate evidence supporting both active and passive proprioception deficits in CAI as compared with controls. According to the latest systematic review and meta-analysis by Xue et al. (2021), CAI-affected ankles had poorer ankle kinesthesia in both inversion and plantarflexion when compared with the contralateral side; and individuals with CAI showed kinesthesia defects and active joint reposition deficits in the frontal plane movement (both inversion and eversion) when compared to the healthy controls. Not until recent years that more attention has been drawn to deficits in cutaneous sensation. Hoch et al. (2012) found that the plantar surface was less sensitive to vibratory tactile stimulation as compared to non-CAI people at the head of the first metatarsal, the base of the fifth metatarsal, and the heel, along the innervation of the branches of the sural and tibial nerves. Burcal and Wikstrom found similar results that people with CAI displayed higher Semmes Weinstein monofilament thresholds at the head of the first metatarsal, base of the fifth metatarsal, and sinus tarsi31. The possible involvement of impaired cutaneous sensation in CAI have led to the recent approach of sensory-targeted intervention in this population.

Deficits in central sensorimotor control in CAI: As described in the previous paragraphs that the classic theory behind the ankle instability has been based on damages of joint receptors and peripheral nerve fibers. However, emerging data has shown that proprioceptive sensory deficits were not enough to explain the neuromuscular deficits in people with CAI, and that more research is needed to determine how CAI influences central sensorimotor control.

Previous studies have shown that in individuals with chronic musculoskeletal dysfunction such as shoulder impingement and low back pain, the integration of corticospinal pathways may be affected, presented as higher active motor threshold, longer cortical silent period, reduced cortical mapping area and shifted center of gravity of the cortical mapping area. Possible impairment of the corticospinal control in CAI has recently been examined in a few studies. While Pietrosimone and Gribble (2012), Shih et al. (2017), and Terada et al. (2022) reported that muscles around the ankle joint had impaired corticospinal excitability (reduced motor-evoked potential of the peroneus longus and soleus muscles), the two systemic reviews with meta analysis did not support these findings and showed that people with or without CAI had similar supraspinal neural excitability. These inconsistencies might be related to the differences in study design, such as testing positions and tasks.

The role of altered central motor system excitability in CAI has yet to reach agreement; and little was known about the effect of CAI on the somatosensory cortex. Common outcome measures to evaluate somatosensory cortical activation use electroencephalography (EEG) to detect electrophysiological signals of excitatory and inhibitory action potentials in various areas of the cortex. Previous studies reported abnormalities of P27 potentials and somatosensory-evoked potentials (SEPs) in people with anterior cruciate ligament (ACL) deficits, indicating somatosensory cortex neuroplasticity following ACL injuries. Only one study has evaluated the somatosensory cortical activation in people with ankle instability, and found no difference in somatosensory cortical activity (event-related desynchronization (ERD) of the upper alpha frequency) between healthy controls and individuals with unstable ankles. With strong evidence showing connections between central sensorimotor deficits and chronic musculoskeletal problems such as low back pain and ACL deficits, we believe that future research is required to understand the role of sensory deficits, particularly the central somatosensory activation in people with CAI and to provide further explanation for the neurophysiological mechanisms for ankle instability.

Restoration of motor performance has been the popular intervention for CAI: From the above review, it is obvious that problems behind chronic ankle instability relate to both sensory and motor systems. However, the majorities of intervention strategies have focused on restoring the defects in motor pathways, including muscle strengthening, neuromuscular training, posture and balance control training. Although many of the studies found positive effects of these motor restoration interventions, the synthesis of evidence only supported partially (limited to moderate level) for the effectiveness of neuromuscular or balance training on muscle performance, postural stability or self-perceived improvement.

Emerging evidence showing effectiveness of sensory-orientated intervention for CAI: With more understanding on the involvement of sensory deficits in CAI, some researchers started to describe intervention methods using primarily sensory inputs, such as planar massage, and joint mobilization. Joint mobilization was found to improve dynamic posture performance including landing kinematics, reaching distances of the Y balance test, ankle mobility, and self-perceived dysfunction questionnaires. Although joint mobilization was proposed to have the effect of "resetting the sensorimotor control", the spinal-reflex and corticospinal excitability of the soleus and peroneus longus were not altered after one session of joint mobilization. In addition, joint mobilization not only provides sensory stimulation but also offers alignment correction for people with CAI. The effectiveness of joint mobilization could have come from improvement in ankle mobility rather than sensory intervention. Several studies have investigated the effect of pure sensory inputs, the plantar massage, in people with CAI and found that plantar massage effectively improved static postural control. However, these studies only measured perceived dysfunction, or functional performance. No neurophysiological mechanism of sensory intervention in CAI has been explored before.

Electrical stimulation as a form of treatment for CAI: Traditionally, neuromuscular stimulation has been used as a form of treatment for various conditions, from peripheral nerve injuries, conditions involving arthrogenic inhibition such as ACL insufficiency or patellofemoral pain, to neurological conditions including stroke or spinal cord injury. A great body of evidence has shown that neuromuscular stimulation is effective in restoring motor functions in these conditions. Another approach of electrical stimulation is to use sensory level of stimulation in attempt to improve sensorimotor control. The rationale is that somatosensory stimulation would enhance cortical plasticity in people post stroke. Pan et al. recruited 12 patients post stroke and assessed the effect of 40 minutes of sensory electrical stimulation, combined with hand rehabilitation program. The changes in sensorimotor control were evaluated using corticomuscular coherence (CMC). After 4 weeks of treatment, the CMC value of the electrical stimulation group is higher than that of the control group, indicating that the cerebral motor cortex and the corresponding muscles have a greater and physiologically meaningful functional connection. Although people with CAI has been found to have benefited from sensory intervention such as plantar massage, no neurophysiological mechanism has been studied. In addition, application of sensory transcutaneous electrical stimulation (TENS) is a relatively risk-free and easy-to-implement modality for rehabilitation. However, no study has investigated the effect and treatment mechanisms of TENS in people with CAI.

Research gap and contribution of the study: Current research evidence supported that people with chronic ankle instability have deficits in peripheral sensorimotor systems and central motor impairments, resulting in defects in sensorimotor control and functional performance. However, little was known about how CAI affects the somatosensory cortical activation. The effects of strength training, neuromuscular control training, posture/balance training has been widely investigated for CAI, and positive effects on neuromuscular control, corticospinal excitability, and functional performance have been found for this group of people. Recently, sensory intervention for CAI has been proposed and its treatment effect on static and dynamic posture control as well as functions were reported. Based on the effectiveness of sensory intervention and posture adaptation strategies shown in individuals with CAI, it is reasonable to speculate that central somatosensory processing might have a role in altered neuromuscular performance and recovery (sensory intervention effect) of CAI. However, these neurophysiological mechanisms have never been studied before.

To address the above issues, we would like to apply for a three-year grant to firstly investigate the effect of CAI on somatosensory cortical activation, corticomuscular coherence, proprioception, cutaneous sensation of the plantar surfaces, and neuromuscular performance. These variables will be compared between 45 young active adults with CAI and 15 controls for the first year study. Secondly, those with CAI will be randomized into three groups, the sensory stimulation group, the sham stimulation group, and the control group. The participants will receive 40 minutes of sensory level of electrical stimulation or sham stimulation or nothing, and the immediate effect will be examined to understand the effect of sensory-level stimulation on neurophysiological mechanisms and neuromuscular performance. Afterwards, the intervention (sensory stimulation with exercise, sham stimulation with exercise, and exercise alone) will be carried out for 5 sessions in two weeks, and the short term intervention effect of additional sensory stimulation will be assessed.

The results of this study will provide a better understanding for sensorimotor control in CAI, and for the effect of sensory stimulation intervention in the population with CAI. The data from this investigation will provide clinicians, trainers, and researchers an excellent basis for the management and injury prevention of CAI among athletes, and for further research in this field of study.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 40 years old
* having at least one ankle sprain experience in the past year with sequelae; or having repeated ankle sprain experience in the past year,
* having a "soft foot" sensation within three months
* score ≤ 27 on the Cumberland Ankle Instability Tool (CAIT)

Exclusion Criteria:

* having a history of lower extremity fracture or surgery, or a history of lower extremity trauma in the past three months
* having experiences of sprained ankles within the previous six weeks
* having pathological joint laxity (positive results on talar tilt test or drawer forward test

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Cortical activation | 5 minutes
  somatosesory evoked potentials and corticomuscular coherence

SECONDARY OUTCOMES:
Proprioception | 10 minutes
  ankle inversion and plantarflexion joint position sense
Two-point discrimination | 10 minutes
  Cutaneous sensation of the plantar surfaces
Range of motion | 5 minutes
  ankle dorsiflexion range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim KM, Ingersoll CD, Hertel J. Altered postural modulation of Hoffmann reflex in the soleus and fibularis longus associated with chronic ankle instability. J Electromyogr Kinesiol. 2012 Dec;22(6):997-1002. doi: 10.1016/j.jelekin.2012.06.002. Epub 2012 Jul 13. PMID 22795679
- [Background] Kim KM, Kim JS, Cruz-Diaz D, Ryu S, Kang M, Taube W. Changes in Spinal and Corticospinal Excitability in Patients with Chronic Ankle Instability: A Systematic Review with Meta-Analysis. J Clin Med. 2019 Jul 16;8(7):1037. doi: 10.3390/jcm8071037. PMID 31315231
- [Background] Suttmiller AMB, McCann RS. Neural excitability of lower extremity musculature in individuals with and without chronic ankle instability: A systematic review and meta-analysis. J Electromyogr Kinesiol. 2020 Aug;53:102436. doi: 10.1016/j.jelekin.2020.102436. Epub 2020 Jun 1. PMID 32505988
- [Background] Wikstrom EA, McKeon PO. Predicting balance improvements following STARS treatments in chronic ankle instability participants. J Sci Med Sport. 2017 Apr;20(4):356-361. doi: 10.1016/j.jsams.2016.09.003. Epub 2016 Sep 20. PMID 27840034
- [Background] Shih YF, Yu HT, Chen WY, Liao KK, Lin HC, Yang YR. The effect of additional joint mobilization on neuromuscular performance in individuals with functional ankle instability. Phys Ther Sport. 2018 Mar;30:22-28. doi: 10.1016/j.ptsp.2017.12.001. Epub 2017 Dec 20. PMID 29310055
- [Background] McKeon PO, Wikstrom EA. Sensory-Targeted Ankle Rehabilitation Strategies for Chronic Ankle Instability. Med Sci Sports Exerc. 2016 May;48(5):776-84. doi: 10.1249/MSS.0000000000000859. PMID 26717498
- [Background] Pan LH, Yang WW, Kao CL, Tsai MW, Wei SH, Fregni F, Chen VC, Chou LW. Effects of 8-week sensory electrical stimulation combined with motor training on EEG-EMG coherence and motor function in individuals with stroke. Sci Rep. 2018 Jun 15;8(1):9217. doi: 10.1038/s41598-018-27553-4. PMID 29907780
- [Background] Kim KM, Croy T, Hertel J, Saliba S. Effects of neuromuscular electrical stimulation after anterior cruciate ligament reconstruction on quadriceps strength, function, and patient-oriented outcomes: a systematic review. J Orthop Sports Phys Ther. 2010 Jul;40(7):383-91. doi: 10.2519/jospt.2010.3184. PMID 20592480
- [Result] Xue X, Ma T, Li Q, Song Y, Hua Y. Chronic ankle instability is associated with proprioception deficits: A systematic review and meta-analysis. J Sport Health Sci. 2021 Mar;10(2):182-191. doi: 10.1016/j.jshs.2020.09.014. Epub 2020 Oct 2. PMID 33017672
- [Result] Needle AR, Lepley AS, Grooms DR. Central Nervous System Adaptation After Ligamentous Injury: a Summary of Theories, Evidence, and Clinical Interpretation. Sports Med. 2017 Jul;47(7):1271-1288. doi: 10.1007/s40279-016-0666-y. PMID 28005191